CLINICAL TRIAL: NCT03789513
Title: Evaluation of Screening Algorithms Based on Self-collection and HPV Testing With Partial Genotyping for the Prevention of Cervical Cancer Among HIV-infected Women in Low-income Countries
Brief Title: Evaluation of Triage Options After HPV Testing for Cervical Cancer Screening Among HIV-infected Women
Acronym: AIMA-CC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Institut de Recherche pour le Developpement (Other Government); International Agency for Research on Cancer (Other); Programme PAC-CI, Site ANRS-MIE de Côte d'Ivoire (Other); University Hospital, Geneva (Other); University of Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ANRS12375 AIMA-CC
Record Dates: First submitted 2018-09-03; First posted 2018-12-28 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: HIV Infections; HPV - Anogenital Human Papilloma Virus Infection
Keywords: HIV infection, HPV infection, cervical cancer, screening algorithms; recurrence
MeSH Terms: conditions — HIV Infections; Papillomavirus Infections; Uterine Cervical Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Triage with different options (Other): All women will have an HPV test, partial genotyping (16/18/45 versus other high-risk HPV [hr-HPV]) and VIA. The different options for triage that will be compared are:
  * Participants hr-HVP+ and VIA+ participants selected for treatment;
  * Participants HPV 16/18/45+ selected for treatment;
  * Participant HPV 16/18/45+ and/or VIA+ selected for treatment;
  Interventions: Diagnostic Test: HPV test with partial genotyping and VIA triage

INTERVENTIONS:
Diagnostic Test: HPV test with partial genotyping and VIA triage — HPV testing with the GenXpert platform VIA Biopsies of VIA+ lesions or random Treatment with thermal ablation of women with precancerous lesions

SUMMARY:
Cervical cancer is the most common cause of cancer and a leading cause of death among HIV-infected women living in resource-limited settings. Although screening for premalignant lesions is an effective way of reducing cervical cancer incidence, its uptake in low-resource settings to date is low. The use of HPV testing for primary screening is currently recommended by many guidelines - including the WHO guidelines for cervical cancer screening in resource-limited settings - because of its greater sensitivity and ease of use compared to other options. However, these WHO guidelines have both highlighted the need to conduct more research on appropriate HPV-based algorithms among HIV-infected women, as immunodeficiency may affect the screening performance. Indeed, HPV infections in HIV-infected women are very common, so there is a need for additional triage to identify women most at risk and there remains considerable uncertainty on the optimal option for such triage. Most of the evidence available comes from HIV-negative populations living in high-resource settings and is not necessarily relevant for low-resource contexts where the epidemiological background is different, women access late to screening and may not have follow up visits, where financial constraints are important and health service resources limited.

Hence, the proposed project aims to provide evidence on the effectiveness and feasibility of HPV-based screening algorithms among HIV-infected women in low-resource settings.

This multicenter cross-sectional study will include 3,000 HIV-infected women (30-49 years old) receiving HAART and followed in Abidjan (Ivory Coast), Bobo-Dioulasso (Burkina Faso) and Phnom Penh (Cambodia).

After self-collection of cervico-vaginal samples, each participant will have an HPV test with partial genotyping primary using the Xpert HPV assay, a real-time PCR assay that provides the possibility of identifying 14 HR-HPV types within one hour. The Xpert HPV test has been chosen because of the wide availability of the Genexpert platform in HIV care centers from resource-limited settings. Furthermore, it can specifically detect HPV-16, 18 and 45, the most carcinogenic HPV types in both HIV-negative and HIV-positive women, separately from other high-risk HPV types. VIA will be another triage option either alone or combined to HPV DNA genotyping.

In addition, participants treated for cervical lesion will be followed over 12 months to assess the risk of post-treatment lesions (CIN2+/HSIL) and to identify associated risk-factors.

ELIGIBILITY:
Inclusion Criteria:

* Women
* HIV-1 infection
* Age 30 to 49 years
* In care for HIV infection, receiving or initiating antiretroviral therapy
* Written informed consent given

Exclusion Criteria:

* HIV-2 infection
* Ongoing pregnancy (evidenced by self-report or clinical examination)
* Previous total hysterectomy
* Severe concomitant disease that, according to the investigators, may contraindicate or compromise participation to the study
* History of cervical cancer screening with treatment for precancerous lesions within the last 12 months

Differed inclusion

* Ongoing heavy menstruation
* Immediate post-partum (<12 weeks post delivery)
* Sign of ongoing genital infection (e.g. mucopurulante discharge)

Ages: 30 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3000 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the triage options | Day 0
  Sensitivity of the triage options to detect CIN2+ and CIN3+ lesions with histology as the reference standard
Specificity of the triage options | Day 0
  Specificity of the triage options to detect CIN2+ and CIN3+ lesions with histology as the reference standard

SECONDARY OUTCOMES:
Positive and negative predictive value (PPV and NPV) of the triage options | Day 0
  PPV and NPV of the triage options to detect CIN2+ and CIN3+ lesions with histology as the reference standard
Positive and negative diagnostic likelihood ratio (DLR) of the triage options | Day 0
  Positive and negative DLR of the triage options to detect CIN2+ and CIN3+ lesions with histology as the reference standard
Acceptability and feasibility | Day 0 and Week 1
  Acceptability and feasibility of the self-sampling, of the different triage options and of the treatment cervical lesions
Prevalence of CIN2+ lesions | Day 0
  Prevalence of CIN2 lesions, overall and by sub-groups defined by age categories, current CD4-cell count, nadir CD4-cell count and treatment history
Prevalence of CIN3+ lesions | Day 0
  Prevalence of CIN3 lesions overall and by sub-groups defined by age categories, current CD4-cell count, nadir CD4-cell count and treatment history
Prevalence of cervical cancer | Day 0
  Prevalence of cervical cancer overall and by sub-groups defined by age categories, current CD4-cell count, nadir CD4-cell count and treatment history
Adverse events | Day 0 and Week 1 up to 24 weeks
  Rate and nature of adverse events and protocol violations
Proportion of the women eligible to HPV screening who were actually screened and treated (if required) | Day 0
  Proportion of the women eligible for the study who were actually screened, treated (if required)
Evaluation of the micro-costing | Day 0 up to Week 26
  Evaluation of the micro-costing of the various components of the screening strategies
Evaluation of post-treatment HPV clearance | Week 24 and 48 post treatment
  Evaluation of the HPV clearance at M6 and M12 after thermal-ablation
Evaluation of post-treatment cervical lesion | Week 48 post treatment
  Evaluation of the proportion of CIN2 and CIN3 at M12 after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Debeaudrap, PhD, Study Director — Ceped UMR 196; Apollinaire Debeaudrap, PhD, Study Director — PACCI - Ivory Coast
Locations (3):
- HIV day care center, Bobo-Dioulasso, Burkina Faso
- Calmette Hospital, Phnom Penh, Cambodia
- CEPREF, Abidjan, Côte d’Ivoire

IPD SHARING:
Plan to Share IPD: No